CLINICAL TRIAL: NCT01201720
Title: Effects on Plasma Exchange on Functional Capacity of Serum Albumin, Circulatory Liver Failure"
Brief Title: Effects on Plasma Exchange on Functional Capacity of Serum Albumin, Circulatory Dysfunction, Renal and Cerebral Function in Cirrhotic Patients With "Acute-on-chronic Liver Failure"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Grifols, S.A. (Industry)
Responsible Party: Sponsor
Organization: Grifols Therapeutics LLC (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IG0905; 2010-021360-15 (EudraCT Number)
Record Dates: First submitted 2010-08-27; First posted 2010-09-15 (Estimated); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Liver Cirrhosis; Liver Failure
Keywords: cirrhosis; cirrhotic patients with acute on chronic liver failure
MeSH Terms: conditions — Liver Cirrhosis; Liver Failure; Fibrosis | interventions — Plasma Exchange; Albumins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Albumin (Other): Albumin solution for infusion 5%. dosage: 43,5 millimole intravenouse use , 6 plasma exchange with albumin in 11 days and administration of polyclonal gamma globulin.6 sessions
  Interventions: Procedure: Plasma exchange with albumin

INTERVENTIONS:
Procedure: Plasma exchange with albumin — Realization of 6 plasma exchange with albumin in 11 days
  Other Names: Albumina grifols 5%

SUMMARY:
The purpose of this study is to evaluate the effects on plasma exchange with 5% albumin on albumin functional capacity, cardiocirculatory, renal and cerebral function in cirrhotic patients with "acute-on-chronic liver failure".

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effects on plasma exchange with 5% albumin on albumin functional capacity, cardiocirculatory, renal and cerebral function in cirrhotic patients with "acute-on-chronic liver failure", renal disfunction, cerebral disfunction ,and inflamtory response

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years old
* Hepatic cirrhosis diagnosed by biopsy or clinical, analytic and ultra sound data.
* acute on chronic liver failure: defined by an acute deterioration in hepatic function produced in 2-4 weeks with jaundice (total serum bilirubin ≥ 5 mg/dl ) and hepatic encephalopathy (≥ grade 2) and/or renal insufficiency (serum creatinine ≥ 2 mg/dl)

Exclusion Criteria:

* Neoplasm disease including hepatocarcinoma which exceed Milan criteria (1 tumour > 5cm, up to 3 tumours <3 cm)
* Active bacterial or fungal infection with hemodynamic instability which require the utilization of vasoactive drugs at moderate dose (>0,5 μg/Kg/min of noradrenaline)
* Structural moderate to severe cardiopathy (Cardiac Index <2l/min/m2)
* Chronic renal insufficiency in treatment with haemodialysis
* Chronic moderate o severe pulmonary disease (maximum expiratory volume in a second <50%)
* Active transplant
* human immunodeficiency virus infection
* Pregnancy or lactation
* Acute respiratory distress syndrome (P02/Fi02< 200mm Hg) or acute lung injury (P02/Fi02< 300mm Hg)
* Hemodynamic instability (>0,5 μg/Kg/min of noradrenaline)
* Bleeding in the digestive tract in the previous 72h to the treatment
* Severe coagulopathy: INR ≥ 3.0 (Quick ≤ 20%) and/or platelets < 30000//mm3
* Extrahepatic cholestasis
* Hepatobiliary surgery in the last 6 months (except laparoscopic Cholecystectomy)
* Concentrations bilirubin ≥ 5mg/dl during the period above 4 weeks previous to inclusion
* Concomitant participation in an other clinical trial
* Drug addiction
* Mental status which does not allow the patient to understand the trial, with the exception of hepatic encephalopathy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-03; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Albumin functional capacity | 10 days
  Albumin binding capacity
Albumin functional capacity | 10 days
  Electron Paramagnetic Resonance Spectroscopy
Albumin functional capacity | 10 days
  Ischemia-modified albumin
Circulatory disfunction | 10 days
  Plasma renin activity
Circulatory disfunction | 10 days
  Plasma concentration of noradrenaline
Circulatory disfunction | 11 days
  Systemic hemodynamic study and portal venous pressure

SECONDARY OUTCOMES:
Plasma concentration of blood urea nitrogen | 1 month
Hepatic encephalopathy graded with the West Haven Criteria | 1 month
Hepatic function parameters | 1 month
  Conventional hepatic function parameters: aspartate transaminase, alanine transaminase, gamma-glutamyl transferase, alkaline phosphatase, total, conjugated and not conjugated serum bilirubin, serum albumin, international normalized ratio (INR) and prothrombin index
Plasma concentration of serum creatinine | 1 month
Plasma concentration of sodium | 1 month
Plasma concentration of potassium | 1 month
Plasma concentration of phosphorus | 1 month
hepatic toxins | 10 days
  Hepatic toxin concentration: biliary acids, aromatic amino acids, ammonium and lactatum.

CONTACTS AND LOCATIONS:
Overall Officials: Vicente Arroyo, MD, Principal Investigator — Hospital Clínic of Barcelona
Locations (1):
- Hospital Clínic of Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Fernandez J, Lozano M, Torres M, Horrillo R, Afonso N, Nunez L, Mestre A, Perez A, Cid J, Costa M, Arroyo V, Paez A. Effect of plasma exchange with albumin replacement on albumin functionality and organ dysfunction in acute-on-chronic liver failure. JHEP Rep. 2024 Jan 22;6(4):101017. doi: 10.1016/j.jhepr.2024.101017. eCollection 2024 Apr. PMID 38544553